CLINICAL TRIAL: NCT05338268
Title: Addressing Loneliness and Substance Use With Telehealth CBT
Brief Title: Substance Use and Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPO 21-074
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders
Keywords: Loneliness; Substance use disorders; social isolation; drug use
MeSH Terms: conditions — Substance-Related Disorders; Social Isolation

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two interventions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessors will not know what condition that the participant was allocated to, nor will the statistician who is one of the co-investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT for Loneliness (Experimental): CBT focused on social relationships and loneliness delivered over the course of 8, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: CBT for Loneliness
- CBT for Substance Use Disorder (Active Comparator): CBT focused on substance use disorders delivered over the course of 8, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: CBT for Substance Use Disorder

INTERVENTIONS:
Behavioral: CBT for Loneliness — CBT focused on social relationships and loneliness delivered over the course of 8, ~45 minute sessions delivered via telehealth.
  Arms: CBT for Loneliness
Behavioral: CBT for Substance Use Disorder — CBT focused on substance use disorders delivered over the course of 8, ~45 minute sessions delivered via telehealth.
  Arms: CBT for Substance Use Disorder

SUMMARY:
Background: Loneliness-a subjective emotional state characterized by the perception of social isolation-is a psychosocial factor that is associated with increased mortality, substance use, and is associated with precipitants of relapse among individuals with substance use disorders (SUD). Importantly, there are effective interventions that can be used to decrease loneliness; however, these have not been tested on Veterans with SUD who are lonely.

Significance/Impact: Individuals with SUD have higher prevalence of loneliness and loneliness exacerbates pain and sleep disturbance, risk factors of relapse. Without effectively intervening on loneliness, Veterans with SUD will continue to be at high risk of relapse and will maintain problems engaging with social support, including healthcare providers-factors critical for recovery. Cognitive-behavioral therapies (CBT) has shown the strongest effects on loneliness, however, there are no interventions that are specifically designed for substance using populations who are lonely. Testing CBT for loneliness and SUD (CBT-L/SUD) has the potential to have a broad impact on addressing a critical, unmet need that commonly affects Veterans with SUD. The investigators approach of national recruitment and telehealth delivery of this intervention highlights how this this study address VHA care priorities including substance use, access to care, and telehealth.

Innovation: There are no studies that have tested a loneliness intervention in Veterans with SUD who are lonely, which may neglect a broader impact on mental and physical health. This study is ideally situated to generate new and important knowledge on the association of loneliness and SUD. This study seeks to address a transdiagnostic factor, which may improve engagement with social support thereby reducing substance use. An additional innovative aspect of this study is recruitment being conducted outside the VHA. This may increase access to care among those Veterans who are especially isolated.

Specific Aims: the investigators aim to: (1) refine the CBT-L/SUD manual by conducting a one-arm trial among Veterans with a SUD who report loneliness (n = 6), (2) randomize participants to receive either CBT-L/SUD (n = 15) or CBT-SUD (n = 15) to assess feasibility and acceptability among Veterans with a SUD who report loneliness.

Methodology: the investigators will elicit feedback on a draft of the CBT-L/SUD manual then conduct a small single-arm trial (n = 6) for further refinement. Specifically, SUD treatment providers and Veterans with SUD will provide feedback on the draft manual, which the research team will integrate to finalize the manual for a small single-arm trial. This trial will allow us to collect feasibility of treatment delivery, and treatment satisfaction and acceptability data to further refine the manual. With the refined manual Veterans with SUD reporting loneliness will be randomized to either CBT-L/SUD (n = 15) or CBT-SUD (n = 15). The investigators will assess: (1) treatment acceptability, (2) participant adherence to treatment, and (3) therapist fidelity. The investigators will also assess outcome measure completion percentage, means and standard deviations, and level of correlation of repeated measurement of primary loneliness outcomes and secondary substance use outcomes.

Implementation/Next Steps: Results from this study will provide critical feasibility and acceptability data to inform an HSR&D Merit Award application to conduct a fully-powered randomized controlled trial. The research team will work with the VA Office of Mental Health and Suicide Prevention and the Substance Use Disorder office of the National Mental Health Program to identify implementation and dissemination efforts. For example, the investigators plan to translate findings into applied practice across various settings (e.g., primary care mental health, rehabilitation treatment programs). Additionally, this intervention may be particularly useful for behavioral telehealth centers that deliver evidence-based interventions to rural and other Veterans who have difficulty accessing VHA care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ages 18+,
* understand English,
* have access to a phone or computer,
* screen positive for an active, at least moderate SUD. SUD include alcohol, marijuana, opioids, cocaine, other psychomotor stimulants (methamphetamine, amphetamines), and sedative/hypnotic/anxiolytic use disorders.
* Participants will need to screen positive for loneliness.

Exclusion Criteria:

* Participant with significant cognitive impairment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisham Ashrafioun, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited through a case finding procedure of VHA medical records.
Pre-assignment Details: The first 6 participants all received CBT for Loneliness after a baseline assessments. For the next 30 participants, participants in both conditions receive a baseline assessment and then were randomized to either CBT for Substance Use Disorders or CBT for Loneliness.
Period: Overall Study
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Started | 20 | 16
Completed | 9 | 5
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- CBT for Loneliness: CBT for social relationships and loneliness delivered over the course of 8, ~45 minute sessions delivered via telehealth.
- CBT for Substance Use Disorder: CBT for substance use disorders delivered over the course of 8, ~45 minute sessions delivered via telehealth.
- Total: Total of all reporting groups
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.45 (14.0) | 39.81 (11.55) | 42.39 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 16 | 12 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Loneliness
Description: Loneliness will be measured using the UCLA Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: Participant flow includes participants from the one-arm trial. Participants reported in the outcomes do not include participants from the one-arm trial because there was not a one-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 8 | 5
score on a scale | -1.38 (17.82) | -5.40 (3.58)

2. Secondary Outcome: Mean Change in Number of Days of Substance Use
Description: Participants will complete a calendar indicating the type and frequency of substance use.
Time Frame: baseline to 1-month post-treatment
Population: Participant flow includes participants from the one-arm trial. Participants reported in the outcomes do not include participants from the one-arm trial because there was not a one-month follow-up. Data missing for one participant in each arm compared to other outcomes of interest.
Measure: Mean (Standard Deviation); unit: percentage of days (used/total)
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 7 | 4
percentage of days (used/total) | -1.79 (3.74) | -1.75 (1.26)

3. Secondary Outcome: Mean Change in Percent Days Abstinent
Description: Participants will complete a calendar indicating the type and frequency of substance use
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of days (abstinent/total)
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 7 | 4
percentage of days (abstinent/total) | 5.95 (12.74) | 5.83 (4.19)

4. Secondary Outcome: Mean Change in Social Interactions
Description: Duke Social Support Index assesses several domains of perceived social support, including social network size, social interaction, social satisfaction, and instrumental social support. Higher scores indicate a higher quality of social interactions. Scores range from 0 to 37.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 8 | 5
units on a scale | .38 (6.05) | 4.00 (1.73)

5. Other Pre Specified Outcome: Mean Change in Depression
Description: Depression will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 8 | 5
units on a scale | -2.00 (6.95) | -2.80 (2.17)

6. Other Pre Specified Outcome: Mean Change in Anxiety
Description: Anxiety will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
Number analyzed (Participants) | 8 | 8
units on a scale | .13 (4.45) | -5.80 (3.11)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up (baseline assessment, post-treatment assessment, 1-month follow-up; 8 intervention session; ~3 months)
Arm/Group | CBT for Loneliness | CBT for Substance Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/16
Other Adverse Events (participants affected / at risk) | 3/20 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT for Loneliness (N=20) | CBT for Substance Use Disorder (N=16)
hospitalization - detoxification (Psychiatric disorders) | 1 (1) | 0 (0)
hospitalization - GI issues (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT for Loneliness (N=20) | CBT for Substance Use Disorder (N=16)
Increased psychiatric distress/substance use (Psychiatric disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT05338268/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT05338268/ICF_000.pdf